CLINICAL TRIAL: NCT00177502
Title: Effect of Exercise on Prevention of Weight Gain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R01HL070257-01A1 (NIH); R01HL070257-01A1 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-09

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

INTERVENTIONS:
Behavioral: behavioral exercise intervention

SUMMARY:
The purpose of this study is to examine the dose-response of exercise on prevention of weight gain in overweight adults.

ELIGIBILITY:
Inclusion Criteria:

1. Female or Male
2. 18-55 years of age
3. BMI = 25-29.9 kg/m2
4. Ability to provide informed consent.
5. Ability to provide consent from their personal physician to participate in this study.

Exclusion Criteria:

1. Reporting regular exercise participation of at least 20 minutes per day on at least 3 days per week during the previous six months. (This study is designed to recruit relatively sedentary adults.)
2. Diabetes, hypothyroidism, or other medical conditions which would affect energy metabolism.
3. Women who are currently pregnant, pregnant within the previous six months, or planning on becoming pregnant within the next 12 months. (Pregnancy during initial screening will be based on self-report and will be included on the detailed medical history that is completed by subjects. However, this will be confirmed with the urine pregnancy test that will be conducted prior to the baseline DEXA.)
4. Non-medicated resting systolic blood pressure >160 mmHg or non-medicated resting diastolic blood pressure >100 mmHg, or taking medication that would affect blood pressure.
5. Taking medication that would affect resting heart rate or the heart rate response during exercise (e.g., beta blockade).
6. Arrhythmia on resting or exercise electrocardiogram that would indicate that vigorous exercise was contraindicated.
7. History of myocardial infarction or valvular disease.
8. History of orthopedic complications that would prevent optimal participation in the exercise component (e.g., heel spurs, severe arthritis).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 294
Dates: Start 2003-01; Study Completion 2006-12

PRIMARY OUTCOMES:
body weight

SECONDARY OUTCOMES:
fitness
physical activity
dietary intake
mediators

CONTACTS AND LOCATIONS:
Overall Officials: John M Jakicic, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Janney CA, Jakicic JM. The influence of exercise and BMI on injuries and illnesses in overweight and obese individuals: a randomized control trial. Int J Behav Nutr Phys Act. 2010 Jan 6;7:1. doi: 10.1186/1479-5868-7-1. PMID 20145731